CLINICAL TRIAL: NCT04812249
Title: Effect of Co-morbidities on the Development of Oral Feeding Ability in Pre-term Infants: a Prospective Study at Neonatology Unit of Assiut University Children Hospital
Brief Title: Effect of Co-morbidities on the Development of Oral Feeding Ability in Pre-term Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khalaf Ali, Assistant Lecturer, Assiut University
Other Study IDs: Oral feeding in preterms
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Feeding; Difficult, Newborn; Pre-Term
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical assessment — Clinical assessment and follow up of oral feeding ability

SUMMARY:
The aim of this study is to investigate the effect of co-morbidities on the timing of the achievement of full oral feeding in a cohort of pre-term infants and to evaluate their mode of feeding and feeding status at the time of hospital discharge.

DETAILED DESCRIPTION:
It is widely acknowledged that pre-term infants frequently experience difficulties in attaining independent oral feeding, thus delaying the achievement of an adequate nutritional status and hospital discharge which - according to the American Academy of Pediatrics- requires the ability to feed exclusively by mouth(1-2) The development of oral feeding ability in pre-term infants is therefore a primary concern for neonatologists.

Because of the immaturity of their body functions and the occurrence of co-morbidities, pre-term infants generally require a period of enteral feeding before they acquire the coordinated sucking ability that allows sufficient milk intake for growth(3) Furthermore, infant sucking skills differ between bottle- and breastfeeding (4), and pre-term infants have been reported to show a weaker and less coordinated suck (5).

Few studies have investigated the timing and effect of co-morbidities on the achievement of independent oral skills. Jadcherla et al. (6) reported that infants born with a gestational age of < 28 weeks showed a significant delay in attaining the transition to oral feeding, but it has also been found that the occurrence of morbidities negatively correlates with postmenstrual age at the time of achieving oral feeding skills (6),(7-8).

ELIGIBILITY:
Inclusion Criteria:

1. A randomised sample of all newborns whose gestational age of < 37 weeks .
2. infants who will be admitted to the NICU of Assiut University Children Hospital between 1 May and 31 October 2021.

Exclusion Criteria:

1. known congenital and/or chromosomal diseases.
2. death during hospitalisation, or transfer to another institution.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns whose gestational age of < 37 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean post-menstrual age in weeks at the time of starting and achieving full oral feeding will be evaluated | Baseline
  Statistical analysis will be made using SPSS version 12 software to assess the outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shafeek, Study Director — Assiut University

REFERENCES:
- [Background] Dodrill P, Donovan T, Cleghorn G, McMahon S, Davies PS. Attainment of early feeding milestones in preterm neonates. J Perinatol. 2008 Aug;28(8):549-55. doi: 10.1038/jp.2008.56. Epub 2008 Jun 26. PMID 18580883
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn. Hospital discharge of the high-risk neonate. Pediatrics. 2008 Nov;122(5):1119-26. doi: 10.1542/peds.2008-2174. PMID 18977994
- [Background] Maggio L, Costa S, Zecca C, Giordano L. Methods of enteral feeding in preterm infants. Early Hum Dev. 2012 May;88 Suppl 2:S31-3. doi: 10.1016/S0378-3782(12)70011-7. PMID 22633510
- [Background] Lau C, Geddes D, Mizuno K, Schaal B. The development of oral feeding skills in infants. Int J Pediatr. 2012;2012:572341. doi: 10.1155/2012/572341. Epub 2012 Nov 5. No abstract available. PMID 23193413
- [Background] Capilouto GJ, Cunningham T, Frederick E, Dupont-Versteegden E, Desai N, Butterfield TA. Comparison of tongue muscle characteristics of preterm and full term infants during nutritive and nonnutritive sucking. Infant Behav Dev. 2014 Aug;37(3):435-45. doi: 10.1016/j.infbeh.2014.05.010. Epub 2014 Jun 20. PMID 24956503
- [Background] Jadcherla SR, Wang M, Vijayapal AS, Leuthner SR. Impact of prematurity and co-morbidities on feeding milestones in neonates: a retrospective study. J Perinatol. 2010 Mar;30(3):201-8. doi: 10.1038/jp.2009.149. Epub 2009 Oct 8. PMID 19812589
- [Background] Van Nostrand SM, Bennett LN, Coraglio VJ, Guo R, Muraskas JK. Factors influencing independent oral feeding in preterm infants. J Neonatal Perinatal Med. 2015 May 18;8(1):15-21. doi: 10.3233/NPM-15814045. PMID 25766199
- [Background] Hwang YS, Ma MC, Tseng YM, Tsai WH. Associations among perinatal factors and age of achievement of full oral feeding in very preterm infants. Pediatr Neonatol. 2013 Oct;54(5):309-14. doi: 10.1016/j.pedneo.2013.03.013. Epub 2013 May 7. PMID 23660538